CLINICAL TRIAL: NCT01244269
Title: Two-phase Randomized Controlled Trial of Low and Moderate Dose Methylphenidate for Non-motor and Postural Symptoms in Parkinson's Disease.
Brief Title: The Effect of Methylphenidate on Non-motor Symptoms and Postural Control in Parkinson's Disease.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate enrolment, protocol too challenging for participants, lack of observable benefit after analysis of 6 patients.
Sponsor: Laval University (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Quebec Memory and Motor Skills Disorders Research Center (Other)
Responsible Party: Principal Investigator, Jaime McDonald, Professeur, Laval University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MPH.NMS.2011
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Methylphenidate; Non motor symptoms; Postural control
MeSH Terms: conditions — Parkinson Disease | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- Methylphenidate 10 (Experimental): Methylphenidate 10mg three times daily for a total of 7 doses.
  Interventions: Drug: Methylphenidate
- Placebo 10 (Placebo Comparator): Placebo capsule three times daily for a total of 7 doses.
  Interventions: Drug: Placebo 10
- Methylpheindate 20 (Experimental): Methylphenidate 20mg three times daily for a total of 7 doses.
  Interventions: Drug: Methylphenidate
- Placebo 20 (Placebo Comparator): Placebo capsule three times daily for a total of 7 doses.
  Interventions: Drug: Placebo 20

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate 10mg tablets will be overencapsulated in gelatin capsules for blinding. Subjects will take 1 capsule three times daily for a total of 7 doses.
  Other Names: Ritalin
  Arms: Methylphenidate 10
Drug: Methylphenidate — Methylphenidate 20mg three times daily for a total of 7 doses.
  Other Names: Ritalin
  Arms: Methylpheindate 20
Drug: Placebo 10 — Blind gelatin capsule three times daily for a total of 7 doses.
  Arms: Placebo 10
Drug: Placebo 20 — Blind gelatin capsule three times daily for a total of 7 doses
  Arms: Placebo 20

SUMMARY:
This project aims to determine if methylphenidate can improve deficits in attention and symptoms of orthostatic hypotension, two common non-motor symptoms, in patients with Parkinson's Disease. This project also seeks to evaluate the effect of methylphenidate on postural control in these patients, a debilitating motor symptom that places patients at an increased risk of falling. This study will build on existing data to support a new indication for the use of methylphenidate in Parkinson's Disease. Using standard and objective evaluations, this study will quantify the effect of methylphenidate at two doses on attention levels, orthostatic hypotension, and measures of postural control. Phase I of the study will compare methylphenidate 10mg three times daily to placebo and Phase II of the study, for those tolerating the lower dose in Phase I, will compare methylphenidate 20mg three times daily to placebo. By incorporating two different doses, the study also seeks to determine if any improvements are dose-related. Secondary endpoints will include safety assessments (adverse event monitoring and vital signs) performed every 30 minutes following supervised drug administration. Visual analog scales will be presented to each participant before treatment and following the final dose of each treatment to assess changes in fatigue. A secondary task will be added to postural tests to assess the influence of cognitive processes. It is hypothesized that methylphenidate will demonstrate a significant beneficial effect on all outcomes. It is projected that objective improvements will be observed following treatment with methylphenidate at both doses (10 and 20mg three time daily) when compared to placebo. It is further hypothesized that the effects will be dose-related and therefore more profound with higher doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stages 2-3 Parkinson's disease as defined by the Hoehn &Yahr staging system (Hoehn &Yahr, 1967).
* Age less than or equal to 75 years.
* Subjects who are willing and able to provide, in writing, informed consent.
* Subjects who are willing and able to be confined to the clinical research unit as required by the protocol and to complete all procedures required on an outpatient basis.

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies and excluding seasonal allergies).
* Subjects with a history of substance abuse or dependence or a positive urine screen for drugs of abuse.
* A history of regular alcohol consumption exceeding 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* Subjects with a documented allergy to methylphenidate or one of the product excipients.
* Subjects with any medical condition affecting drug absorption (e.g. gastrectomy).
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Use of a monoamine oxidase inhibitor or other interacting medication within the preceding 14 days or 5 half-lives (whichever is longer).
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Conners' Continuous Performance Test-II score | Baseline, 2 hours following first dose, 2 hours following last dose
Orthostatic drop - blood pressure in mmHg | Baseline, 2 hours following first dose, 2 hours following last dose
  Blood pressure will be measured following 5 minutes of rest in a lying position and again 1, 3, and 5 minutes after rising to a standing position. The orthostatic drop will be calculated by subtracting the blood pressures recorded at each time interval(1, 3, and 5 minutes after standing) from the blood pressure recorded in a lying position.
Average speed of center of pressure oscillations | Baseline, 2 hours following first dose, 2 hours following last dose
  As recorded using dynamic posturography (Sensory Organization Test).
Total area of center of pressure oscillations | Baseline, 2 hours following first dose, 2 hours following last dose
  As recorded using dynamic posturography (Sensory Organization Test).

SECONDARY OUTCOMES:
Visual analog fatigue scale scores | Baseline, 2 hours following last dose
Blood pressure (mmHg) | Baseline, 30, 60, and 90 minutes following first and final dose of study medication
Heart rate | Basesline, 30, 60, and 90 minutes following first and final dose of study medication
Number of errors recorded for 'Backward Digit Span' task | Baseline, 2 hours following first dose, 2 hours following final dose
  Following administration of the Backward Digit Span assessment of the Wechsler Adult Intelligence Scale to control for individual capacities, each subject will be provided with a string of digits before the onset of 50% of the trials in the postural test. Subjects will be required to memorize the string of digits in reverse and repeat them at the end of the trial. Errors will be quantified as either errors of insertion, deletion, or order.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Corbeil, PhD, Study Director — Laval University; Jaime McDonald, BScPhm, Study Director — Laval University; Emmanuelle Pourcher, MD, Principal Investigator — Québec Memory and Motor Skills Disorders Research Center
Locations (2):
- Canada (2):
  - Québec Memory and Motor Skills Disorders Research Center, Québec, Quebec
  - Laval University, Québec, Quebec